CLINICAL TRIAL: NCT06418412
Title: A Pan-Asian Clinical Database of EGFR Exon 20 Insertion Mutated Non-small Cell Lung Cancer (NSCLC)
Brief Title: A Pan-Asian Clinical Database of EGFR Exon 20 Insertion Mutated NSCLC
Status: Recruiting | Type: Observational
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: ATORG006
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Advanced EGFR Exon 20 Insertion Mutated Non-Small Cell Lung Cancer
Keywords: EGFR EXON20 insertion; NSCLC (Non small cell lung cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There are limited in depth studies on the epidemiology and clinical management of EGFR exon 20 insertion mutated NSCLC in Asia. In addition, there is preliminary data suggesting the exact location of the insertion and variant may influence the response and efficacy to novel EGFR targeted therapies.

This study aims to fill this knowledge gap, by comprehensively characterising the epidemiology and clinical outcomes of Asian advanced EGFR exon 20 insertion mutated NSCLC patients.

DETAILED DESCRIPTION:
This study will be a multi-center observational study and will enroll patients with advanced EGFR exon 20 insertion mutated NSCLC.

The study will include patients recruited from countries across Asia, including sites in, but not limited to - Hong Kong, Korea, Singapore, Taiwan and Thailand. There will be approximately 20-30 sites recruiting for the study. In Singapore, sites may include National Cancer Centre Singapore (NCCS), National University Hospital (NUH) and Tan Tock Seng Hospital (TTSH).

Approximately 600 patients will be enrolled retrospectively.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed advanced NSCLC
2. Positive testing result from any locally approved test (including but not limited to RT-PCR, Cobas and NGS) for EGFR exon 20 insertion mutation
3. Diagnosis date from 1 Jan 2013 to 31 Dec 2024 (to allow for minimum 12 months of follow-up clinical and treatment outcome data)
4. Male or female adults, age as defined by local regulations

Exclusion Criteria:

1. Patients without an EGFR exon 20 insertion mutation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced EGFR exon 20 insertion mutated NSCLC.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 10 years.
  Time from diagnosis to death.
Duration of therapy (DOT) | Up to 10 years.
  Time from start of treatment regimen to end of treatment regimen.
Real-world progression-free survival (PFS) | Up to 10 years.
  Time from start of treatment regimen to disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron C. Tan, MBBS, PhD, Study Chair — National Cancer Centre, Singapore; Daniel SW Tan, BSc, MBBS, PhD, Study Chair — National Cancer Centre, Singapore; Dong-Wan Kim, MD, MS, PhD, Study Chair — Seoul National University Hospital; Jin-Yuan Shih, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (3):
- National Cancer Centre, Singapore, Singapore, Singapore
- Seoul National University Hospital, Seoul, South Korea
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No